CLINICAL TRIAL: NCT06271512
Title: A Safety and Effectiveness Registry Study of Patients with Β-Thalassemia Treated with Betibeglogene Autotemcel (the Glostar Registry)
Brief Title: A Study of Participants with Β-Thalassemia Treated with Betibeglogene Autotemcel
Status: Recruiting | Type: Observational
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Collaborators: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Other Study IDs: REG-501
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — Bone marrow and whole blood collected at the time of bone marrow sample collection will be stored centrally to facilitate subsequent exploratory analyses that may include gene/genomic expression studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Participants with β-thalassemia treated with beti-cel in the post-marketing setting will be followed in this registry study for up to 15 years after infusion with beti-cel to collect real-world longitudinal data.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
The main aim of this study is to collect real-world longitudinal data on participants with β-thalassemia treated with betibeglogene autotemcel (beti-cel) in the post marketing setting. To assess the long-term safety, including the risk of newly diagnosed malignancies, after treatment with beti-cel and evaluate the long-term effectiveness of treatment with beti-cel.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be treated with beti-cel in the post marketing setting at a center in the US that participates in the Registry.
* Participant must sign an informed consent and/or assent prior to enrollment as required under applicable laws and regulations.
* Participant must have signed an informed consent and/or assent permitting data to be shared with Center for International Blood and Marrow Transplant Research (CIBMTR).
* Participant must be followed by a hematologist based in the US.

Exclusion Criteria:

- There are no exclusion criteria for Registry participation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with β-thalassemia treated with beti-cel in the post marketing setting at a center in the United States (US) that participates in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2043-12 (Estimated); Study Completion 2043-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who Experience Each Individual Adverse Events of Interest (AEIs) | Through 15 years post-beti-cel infusion
  The Sponsor considers the following events to be AEIs (which should be reported as a medically significant Serious Adverse Event [SAE]):
  * Any newly diagnosed malignancy
  * Neutrophil engraftment failure: defined as healthcare provider (HCP) decision to administer back-up cells or subsequent hematopoietic stem cell transplantation (HSCT) due to neutrophil recovery failure
  * Newly acquired human immunodeficiency virus-1 (HIV-1), HIV-2 infection and human t-lymphotropic virus (HTLV) infection
  * Any newly diagnosed autoimmune disorder
  * Any hepatic veno-occlusive disease (VOD)
  * Any clinically significant bleeding events.

SECONDARY OUTCOMES:
Number of Participants with Serious Adverse Events (SAEs) | Through 15 years post-beti-cel infusion
Number of Participants with beti-cel related AEs | Through 15 years post-beti-cel infusion
Event-Free Survival | Through 15 years post-beti-cel infusion
Percentage of Participants Achieving Transfusion Independence | Through 15 years post-beti-cel infusion

CONTACTS AND LOCATIONS:
Overall Officials: Himal Lal Thakar, MD, Study Director — bluebird bio, Inc.
Locations (6):
- United States (6):
  - UCSF Benioff Children's Hospitals, Oakland, California
  - Stanford University, Palo Alto, California
  - University of Minnesota, Minneapolis, Minnesota
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
bluebird bio is committed to transparency. Appropriately de-identified participant-level datasets and supporting documents may be shared (if bluebird bio is contractually permitted to do so) following completion of this study, completion of all applicable regulatory submissions and consistent with criteria established by bluebird bio, our collaborators and/or industry best practices to protect confidential information and maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.